CLINICAL TRIAL: NCT03230656
Title: Cognitive-Communication Screening and Early Therapy for Adults With Concussion/Mild Traumatic Brain Injury
Brief Title: Cognitive-Communication Screening and Early Therapy for Adults With Mild TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Emi Isaki, Associate Professor, Northern Arizona University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 1003140; 1R15DC015338-01A1 (NIH)
Record Dates: First submitted 2017-07-25; First posted 2017-07-26 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Concussion; Mild Traumatic Brain Injury; Cognitive Communication Disorder
MeSH Terms: conditions — Brain Concussion | interventions — Secondary Prevention

STUDY DESIGN:
Intervention Model Description: Each participant diagnosed with concussion/mild traumatic brain injury will be screened for cognitive and communication abilities at two weeks post-injury and then four weeks post-injury. Standardized scores of the screening measures will identify subjects that are below one standard deviation below the mean. Subjects that continue to exhibit deficits after one month will be randomly placed into an early cognitive-communication therapy group (one month post-injury) or waitlist control group who receive therapy two month post-injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early therapy 1 month post-injury (Experimental): Early cognitive-communication therapy 1 month post-injury:
  * working memory strategies
  * executive function program
  * divided attention program
  * environmental changes
  * identification of problematic cognitive-communication situations
  Interventions: Other: Early cognitive-communication therapy
- Waitlist therapy 2 months post-injury (Active Comparator): Waitlist early cognitive-communication therapy 2 months post injury:
  - Same cognitive-communication therapy is administered
  Interventions: Other: Early cognitive-communication therapy

INTERVENTIONS:
Other: Early cognitive-communication therapy
  Other Names: Early therapy 1 month post-injury; Waitlist therapy 2 months post-injury

SUMMARY:
Approximately 15-20% of patients diagnosed with a concussion/mild traumatic brain injury (mTBI) have persistent symptoms that continue up to six months or longer. Typical problems identified by these patients include difficulty with memory, multi-tasking, the ability to complete tasks quickly, and higher executive functions (e.g., inhibition, initiation, insight, motivation) (Belanger & Vanderploeg, 2005; Mott, McConnon, & Rieger, 2012, Rabinowitz & Levin, 2014). If these symptoms persist they can not only affect thinking, but also communication abilities (e.g., verbal and nonverbal interactions, reading, and writing) (ASHA, 2007). Therefore, it is hypothesized that screening measures that evaluate both thinking and communication can better identify individuals at-risk for persistent symptoms at two week and four weeks post-injury. Also, if cognitive-communication therapy was administered earlier post-injury, then outcomes related to return to daily activities, work, and/or the academic setting could possibly change. This study intends to investigate the use of cognitive and communication screening measures for the identification of persistent symptoms and the provision of early cognitive-communication therapy if problems persist.

DETAILED DESCRIPTION:
Approximately 15-20% of patients with concussion/mild traumatic brain injury (mTBI) have persistent cognitive symptoms up to six months or longer. Problems with working memory, divided attention, processing speed, and executive function are common (Belanger & Vanderploeg, 2005; Mott, McConnon, & Rieger, 2012, Rabinowitz & Levin, 2014). Patients often report how these problems negatively impact daily communication. Although neurocognitive tests are frequently used to identify patients at-risk for persistent symptoms, perhaps tests that not only assess cognition, but also communication would be better at identifying more functional deficits. Patients at-risk for persistent symptoms could then begin therapy earlier to address problems affecting work, school, or everyday activities. Speech-language pathologists are uniquely qualified to evaluate and treat patients with concussion/mTBI and cognitive-communication disorders (ASHA, 2005; Cicerone, et al.; Cornis-Pop et al., 2012). Cognitive-communication is the relationship between cognition and its influence on verbal and nonverbal communication, reading, and writing (ASHA, 2007). At this time, practice guidelines are emerging for cognitive-communication intervention related to concussion/mTBI (Cornis-Pop et al., 2012), yet there is still much research to be done. Typically, in recovery following a concussion/mTBI, patients are referred for cognitive-communication intervention if they are failing or struggling at work, school, or in daily activities. Some patients will not be seen for up to six months based on the assumption by healthcare professionals that most persistent cognitive and communication symptoms will resolve on their own. The wait period before referral for additional services is currently being investigated in the literature. Additionally, therapy for cognitive-communication will only be provided if patients report difficulties to their physicians and are referred for services. If services are not sought out, problems in cognitive-communication will go unrecognized as being a result of the concussion/mTBI.

The specific aims of this study are: 1) Determine if screening measures that evaluate symptoms of concussion/mTBI frequently used by speech-language pathologists administered two and four weeks post-injury will be able to predict individuals at-risk for persistent cognitive and communication symptoms, and 2) Will an early treatment group with persistent cognitive-communication deficits one month after injury differ in pre- and post-therapy functional outcome measure scores as compared to a delayed therapy group beginning services at two months post-injury?

Significance: Results of this study will increase the understanding in the use of cognitive and communication screening measures frequently administered by speech-language pathologists to identify patients at-risk for persistent symptoms related to concussion/mTBI and provide information about the outcomes of cognitive-communication intervention delivered early in recovery.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with concussion/mTBI by ER physician
* speak English as the primary language
* have functional hearing and vision to take the screening measures
* have no prior history of a TBI requiring hospitalization and/or rehabilitation
* have no history of other neurological or psychological diagnoses that would prevent the completion of the screening measures
* mild to moderate hearing loss with aided amplification
* reading glasses to correct their vision
* bilingual subjects whose primary language is English will be included

Exclusion Criteria:

* do not live in Flagstaff, AZ or the surrounding area making them unavailable for follow-up screening or therapy
* English is not spoken as the primary language
* have severe hearing loss or vision problems which cannot be corrected with hearing aids or glasses
* prior history of a traumatic brain injury requiring hospitalization and/or rehabilitation
* history of other neurological or psychological diagnoses preventing the completion of the screening sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
SCAN-A Competing Sentences Subtest | 20 minutes
  Assesses working memory, divided attention, and verbal language
FAVRES Sequencing subtest | 20 minutes
  Evaluates executive function, verbal language, reading, and writing,
WJ-III Tests of Cognitive Abilities Matching subtest | 3 minutes
  Evaluates speed of processing
RBMT-3 Story Immediate and Delayed Recall | 15
  Assesses working memory and verbal language

SECONDARY OUTCOMES:
Functional outcome measure | 40 minutes
  Same outcome measure will be used to determine functional abilities pre- and post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Emi Isaki, Ph.D., Principal Investigator — Northern Arizona University
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to researchers outside of the current study. Results related to the study will be disseminated in future presentations and publications.

REFERENCES:
- [Background] Belanger HG, Vanderploeg RD. The neuropsychological impact of sports-related concussion: a meta-analysis. J Int Neuropsychol Soc. 2005 Jul;11(4):345-57. doi: 10.1017/s1355617705050411. PMID 16209414
- [Background] Mott TF, McConnon ML, Rieger BP. Subacute to chronic mild traumatic brain injury. Am Fam Physician. 2012 Dec 1;86(11):1045-51. PMID 23198672
- [Background] Rabinowitz AR, Levin HS. Cognitive sequelae of traumatic brain injury. Psychiatr Clin North Am. 2014 Mar;37(1):1-11. doi: 10.1016/j.psc.2013.11.004. Epub 2014 Jan 14. PMID 24529420
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Cornis-Pop M, Mashima PA, Roth CR, MacLennan DL, Picon LM, Hammond CS, Goo-Yoshino S, Isaki E, Singson M, Frank EM. Guest editorial: Cognitive-communication rehabilitation for combat-related mild traumatic brain injury. J Rehabil Res Dev. 2012;49(7):xi-xxxii. doi: 10.1682/jrrd.2012.03.0048. No abstract available. PMID 23341288
- See also: Roles of speech-language pathologists in the identification, diagnosis, and treatment of individuals with cognitive-communication disorders [Position Statement] — http://www.asha.org/policy
- See also: Scope of practice in speech-language pathology [Scope of Practice] — http://www.asha.org/policy

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT03230656/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03230656/ICF_001.pdf